CLINICAL TRIAL: NCT04836039
Title: Evaluation of Rehabilitation Experiences of Physiotherapists in Covid-19 Outbreak
Brief Title: Rehabilitation Experiences of Physiotherapists in Covid-19 Outbreak
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pınar Ciddi, Assistant Professor, Medipol University
Other Study IDs: E-10840098-772.02-2682
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Physical Therapy
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapists: Individuals between the ages of 22-65 who continue to work as a self-employed or employee physiotherapist.
  Interventions: Other: A questionnaire and scales.

INTERVENTIONS:
Other: A questionnaire and scales. — Participants will be evaluated by applying a questionnaire and scales created by the researcher physiotherapists based on the researches and examples in the literature.

SUMMARY:
The aim of this study is to evaluate the process experienced by physiotherapists while providing rehabilitation services during the epidemic and to investigate the procedures adopted by physiotherapists who are currently working. In addition, by analyzing the effects of both the pandemic and the clinical and educational organizations in the Physiotherapy and Rehabilitation Clinics where physiotherapists were working during the COVID-19 epidemic, the needs arising after the pandemic can be reported. Assessments will be carried out by researcher physiotherapists through a questionnaire based on research and examples in the literature, and scales measuring anxiety, depression and stress levels. The measurement tool will be the online survey application.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the process experienced by physiotherapists while providing rehabilitation services during the epidemic and to investigate the procedures adopted by physiotherapists who are currently working.

In addition, by analyzing the effects of both the pandemic and the clinical and educational organizations in the Physiotherapy and Rehabilitation Clinics where physiotherapists were working during the COVID-19 epidemic, the needs arising after the pandemic can be reported.

Assessments will be carried out by researcher physiotherapists through a questionnaire based on research and examples in the literature, and scales measuring anxiety, depression and stress levels. The measurement tool will be the online survey application.

Data collection is planned to take place in February-March 2021.

Surveys will be distributed via WhatsApp, e-mail, social media links. This questionnaire was sent to 3 physiotherapists and subjected to a pre-test. This questionnaire is about the following situations and contains 37 questions:

Information on employment status: In this section, physiotherapists' name-surname, gender, age, professional practice experience (years), generally applied physiotherapy subgroup (more than one can be selected), whether they are self-employed or employees, and the status of performing face-to-face clinical practices will be questioned. If so, it will be questioned which protection measures have been applied.

Information about tele-rehabilitation practices: In this section, it will be questioned whether physiotherapists start to follow their patients remotely, if they are, in what way they do it, whether the number of weekly sessions continues, and whether the amount collected is the same as the face-to-face amount.

General information about COVID 19 rehabilitation: In this section, did the departments where physiotherapists work returned to COVID 19 services, did they work in COVID 19 units, rehabilitation approaches in COVID 19 patients, protocol and / or guidelines on exercises for rehabilitation management and treatment of COVID 19 patients. material development / implementation status will be questioned.

The impact of the pandemic on the health and teaching activities of physiotherapists and the sustainability of clinical / thesis studies during this period will be questioned.

Finally, the CES Depression Scale (Center for Epidemiologic Studies Depression Scale, CES-D) will be used to determine depression level, the Generalized Anxiety Disorder 7 (GAD-7) Test will be used to evaluate generalized anxiety level, Perceived Stress Scale (PSS) will be used to determine stress level.

ELIGIBILITY:
Inclusion Criteria:

Individuals between the ages of 22-65 who continue to work as a self-employed or employee physiotherapist.

Exclusion Criteria:

Not meeting the inclusion criteria

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 22-65 who continue to work as a self-employed or employee physiotherapist.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
A questionnaire created by research physiotherapists based on researches and examples in the literature. | The evaluation will take place in one interview (the interview will take 30 minutes)
  Participants will be evaluated by applying a questionnaire and scales created by the researcher physiotherapists based on the researches and examples in the literature.

SECONDARY OUTCOMES:
Assessment of depression level with Center for Epidemiologic Studies Depression Scale | The evaluation will take place in one interview (the interview will take 30 minutes)
  The Center for Epidemiologic Studies Depression Scale will be used to determine depression level. The scale consists of 20 questions in the form of a self-report that measure the emotional state of the person in depression, perceptions and behaviors towards depression. 4-point Likert type questionnaire with 0-60 points range is encoded in 0-3 points range.
Assessment of anxiety level with Generalized Anxiety Disorder 7 Test | The evaluation will take place in one interview (the interview will take 30 minutes)
  The Generalized Anxiety Disorder 7 test will be used to determine anxiety level. It is a 7-item four-point Likert (0 = none, 1 = many days, 2 = more than half of the days, 3 = almost every day), which evaluates the experiences asked in the scale items in the last 2 weeks. The total scores obtained from the scale are 5, 10, and 15 cut-off points for mild, moderate, and severe anxiety, respectively.
Assessment of stress level with Perceived Stress Scale | The evaluation will take place in one interview (the interview will take 30 minutes)
  Perceived Stress Scale will be used to determine stress level. Participants rate how often their lives were seen as unpredictable, uncontrollable, and overly intense during the previous month on the 5-point Likert scale (0 = Never, 4 = Very often). Total scores range from 0 to 40, with higher scores indicating a higher perceived stress level.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, asAss. Prof., Study Chair — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)